CLINICAL TRIAL: NCT02471508
Title: An Innovative Body-Mapping Tank Top Equipped With Biofeedback System for Adolescents With Early Scoliosis
Brief Title: Safety and Efficacy of Body-mapping Tank Top Equipped With Biofeedback System for Adolescent With Early Scoliosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Joanne Yip, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITS/283/13
Record Dates: First submitted 2015-06-11; First posted 2015-06-15 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Adolescent Idiopathic Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tank top with biofeedback system (Experimental): The design of biofeedback tank-top will incorporate sensors to record and monitor the posture of the wearer in real time basis. Alerts will be emitted to the wearer once "poor" posture is detected. The tank-top will be designed to fit the wearer's body and allow the sensor to be placed securely at the targeted position along the spine to minimize the noise from other factors than the wearers' posture and yet comfortable for long-term wearing.
  Interventions: Device: Body-mapping Tank-top Embedded with Biofeedback System

INTERVENTIONS:
Device: Body-mapping Tank-top Embedded with Biofeedback System — In this study, the eligible subjects will be given tailor-made tank-top embedded with biofeedback system to wear it 8 hours daily. Monitor, observation and additional posture training sessions will be provided during the 6 months wearing period. The effectiveness of the biofeedback tank-top will be evaluated by pre-and post- treatment ultrasonic imaging device (measuring the angle of the spine) and electromyography muscle signal

SUMMARY:
Adolescent idiopathic scoliosis (AIS) is a prevalent disease that caused a lateral curvature on spine. Spine curvature increases in youths as puberty progresses. The recommended treatment for AIS is different depends on the spine deformity condition. For mild scoliosis (Cobb's angle ≤ 20°), only periodic observation is suggested. For scoliosis cases that the Cobb's angle ≤ 40°, a rigid brace treatment is recommended. A rigid brace that made by rigid plastic material restrict nearly all movements of the wearers, which caused irritation. Flexible brace is an alternative option, however, the efficiency of such treatment is questionable in terms of controlling the spine curvature progression.

Biofeedback has proven to be effective for a number of physical, psychological and psychophysical problems. The basic aim of biofeedback therapy is to support a patient in realizing his/her self-ability to control specific psychophysiological processes.

In this study, a biofeedback embedded tank-top with a specialized design for adolescents as a treatment option for AIS patients by monitoring the daily posture of the wearers.

DETAILED DESCRIPTION:
This project aims to combine the clinical experience with textiles and biofeedback mechanism to research and develop a biofeedback embedded tank-top for AIS. As a result, this will reduce the future likelihood of brace wear or surgery.

In this study, the eligible subjects will be given tailor-made biofeedback tank-top to wear it 8 hours daily. Monitor, observation and additional posture training sessions will be provided during the 6 months wearing period. The effectiveness of the biofeedback tank-top will be evaluated by pre-and post- treatment ultrasonic imaging device (for measuring the angle of the spine), electromyography muscle signal assessment and clinical photographs assessment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 10 to 13 years
* Diagnosis of AIS in early stage
* Primary Cobb angle between 10 -20 degrees
* Pre-menarche or post- menarche by no more than 1 year
* Ability to read and understand English or Chinese
* At high risk for curve progression
* Skeletally immature (Risser grade 0,1 or 2)
* Physical and mental ability to adhere to functional intimate apparel protocol

Exclusion Criteria:

* Contraindications for x-ray exposure
* Diagnosis of other musculoskeletal or developmental illness that might be responsible for the spinal curvature
* History of previous surgical or orthotic treatment for AIS
* Contraindications for pulmonary and/ or exercise tests
* Psychiatric disorders
* Recent trauma
* Recent traumatic (emotional) event

Ages: 10 Years to 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Progression of the spinal curve | From baseline to 6 months
  No progression of the spinal curve (evaluated by pre-and post- treatment ultrasonic imaging device)

SECONDARY OUTCOMES:
Progression of the spinal curve | From baseline to 6 months
  The progression of the spinal curve within control (increase spinal angle < 5 degrees)
Posture improvement | From baseline to 6 months
  Improvement of posture by clinical photographs assessment and electromyography muscle signal

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, China